CLINICAL TRIAL: NCT05912673
Title: Renal Doppler in Detection of Steroid Resistance in Pediatric Patients With Idiopathic Nephrotic Syndrome
Brief Title: Renal Doppler in Pediatric Patients With Idiopathic Nephrotic Syndrome
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sara Mabrouk Elghoul, Tanta, Stadium Street, Tanta University
Other Study IDs: 36264PR25/1/23
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Nephrotic Syndrome
Keywords: renal doppler; nephrotic syndrome; steroid resistance
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: renal doppler — Toshiba Aplio ultrasound machine and renal resistive index will be measured (peak systolic velocity- end diastolic velocity/ peak systolic velocity

SUMMARY:
The use of the renal resistive index in pediatric patient with idiopathic nephrotic syndrome to detect steroid resistance and to use it as a prognostic instrument of the progression of the disease.

DETAILED DESCRIPTION:
Renal Doppler will be done for all children in supine and lateral positions using Toshiba Aplio ultrasound machine and renal resistive index will be measured (peak systolic velocity- end diastolic velocity/ peak systolic velocity) at diagnosis, after one month, 3 months and 6months, in which these values will be obtained by the ultrasound machine based on the computer algorithm. Also the kidneys will be scanned firstly for length, width, cortical thickness and echogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with primary nephrotic syndrome aged from 1 to 18 years

Exclusion Criteria:

* - Patients with congenital nephrotic syndrome.
* Patients with secondary causes of nephrotic syndrome.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 60 children and adolescents with nephrotic syndrome who will be diagnosed and followed at our nephrology Unit and Clinic at TUH during the period of the study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
detection of steroid resistance in pediatric patients with idiopathic nephrotic syndrome | 6 weeks
  measurement of renal resistive index and detection of steroid sensitivity

SECONDARY OUTCOMES:
progression of nephrotic syndrome | six months
  frequent measurement of renal resistive index and using it as prognostic factor

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mabrouk Mohamed Elghoul, MD, Principal Investigator — Tanta University
Locations (1):
- Sara Mabrouk Mohamed Elghoul, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No